CLINICAL TRIAL: NCT05630781
Title: Orexin's Role in The Neurobiology of Substance Use Disorder
Brief Title: Orexin s Role in the Neurobiology of Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10001066; 001066-DA
Record Dates: First submitted 2022-11-24; First posted 2022-11-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01-23

CONDITIONS: Nicotine Dependence
Keywords: Orexin Antagonish; fMRI; Substance Use Disorder; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders | interventions — suvorexant; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): 80 Volunteers who are between the ages of 18-60 and are non-smokers/vapers. 1. Baseline visit with 1 fMRI scans pre- and post-20mg methylphenidate, 4 acute drug administration (6-14 days in randomized order: 1. Placebo + placebo; 2. 20mg suvorexant + Placebo; 3. Placebo + 40mg methylphenidate; 4. 20 mg suvorexant + 40mg methylphenidate max)
  Interventions: Drug: Belsomra; Drug: Placebo; Drug: Methylphenidate
- Nicotine Dependence Arm (Experimental): 140 Volunteers who are between the ages of 18-60 and are daily smokers/vapers. Suvorexant at 10 mg single dose, and Suvorexant at 10 mg daily for approximately 7 days.
  Interventions: Drug: Belsomra; Drug: Placebo

INTERVENTIONS:
Drug: Belsomra — randomized, double-blind, placebo-controlled crossover design study: Participants will undergo a baseline scan followed by 2 acute drug administration scans where suvorexant or placebo is administered in a randomized manner where both the participant and study staff administering drug are blind. Following the second acute scan, participants will continue with the drug they received at Scan 2 for approximately 7 days. After the first chronic scan, participants will switch to the other drug for an additional approximately 7 days and then scanned a final time.
Drug: Placebo — comparator taken for approximately 10 days
Drug: Methylphenidate — Control Arm: Baseline visit with 2 fMRI scans pre- and post-20mg methylphenidate, 4 acute drug administration (6-14 days in randomized order: 1. Placebo + placebo; 2. 20mg suvorexant + Placebo; 3. Placebo + 40mg methylphenidate; 4. 20 mg suvorexant + 40mg methylphenidate max)
  Arms: Control Arm

SUMMARY:
Study Description:

Despite the availability of pharmacotherapy for some substance use disorders, relapse vulnerability is still a significant issue. This suggests medications with alternative mechanisms of action should be explored to address this unmet need. Substantial preclinical research indicates that orexin antagonism blunts the internally and externally triggered motivation to attain abused substances. This research project will translate these preclinical findings into the clinical domain by administering the FDA approved orexin antagonist, suvorexant, to those with a substance use disorder. Suvorexant s ability to blunt neurobiological correlates of substance misuse will be assessed. This will be assessed following acute and repeated drug administration. Baseline individual differences will be considered to determine whether neurobiological variance influences suvorexant s impact in those with nicotine dependence. In an independent arm, the interaction between suvorexant and a dopamine agonist (methylphenidate) on cognitive function will be assessed in non-smoking individuals.

Objectives:

The objective is to determine the acute and chronic impact of the orexin antagonist, suvorexant, on neurobiological and behavioral factors linked with substance use disorders. Whether such effects are mediated by baseline characteristics will be tested. Given suvorexant is an FDA approved treatment for insomnia, sleep will be evaluated as well in the nicotine dependent arm.

Endpoints:

In nicotine-dependent individuals, suvorexant s impact on brain function will be assessed several ways by evaluating: 1) resting function, 2) reactivity to drug cues, 3) reactivity to non-drug related cognitive tasks. Sleep and nicotine use will be measured throughout the study period. In those without nicotine-dependence, the impact of suvorexant and the interaction of acute methylphenidate and suvorexant on brain function will be assessed. This arm will provide insight into how suvorexant impacts reward/cognition as well as impacts the pharmacological influence of methylphenidate on those same measures.

Study Population:<TAB>

Nicotine dependence arm:140 subjects; Volunteers who are between the ages of 18-60 and are daily smokers/vapers.

Control arm: 80 subjects; Volunteers who are between the ages of 18-60 and are non-smokers/vapers

This study will be conducted at the NIDA-IRP, Biomedical Research Center, in Baltimore, MD.

Description of Study Intervention:

Nicotine dependence arm: Suvorexant at 10 mg single dose, and Suvorexant at 10 mg daily for approximately 7 days.

Control arm: 1. Tolerability visit with one MRI scan post-20mg methylphenidate, 4 acute drug administration (6-14 days in randomized order: 1. Placebo + placebo; 2. 20mg suvorexant + Placebo; 3. Placebo + 40mg methylphenidate; 4. 20 mg suvorexant + 40mg methylphenidate max)

Study Duration:

5 years

Participant Duration:

1-2 months

DETAILED DESCRIPTION:
Study Description:

Despite the availability of pharmacotherapy for some substance use disorders, relapse vulnerability is still a significant issue. This suggests medications with alternative mechanisms of action should be explored to address this unmet need. Substantial preclinical research indicates that orexin antagonism blunts the internally and externally triggered motivation to attain abused substances. This research project will translate these preclinical findings into the clinical domain by administering the FDA approved orexin antagonist, suvorexant, to those with a substance use disorder. Suvorexant's ability to blunt neurobiological correlates of substance misuse will be assessed. This will be assessed following acute and repeated drug administration. Baseline individual differences will be considered to determine whether neurobiological variance influences suvorexant's impact in those with nicotine dependence. In an independent arm, the interaction between suvorexant and a dopamine agonist (methylphenidate) on cognitive function will be assessed in non-smoking individuals.

Objectives:

The objective is to determine the acute and chronic impact of the orexin antagonist, suvorexant, on neurobiological and behavioral factors linked with substance use disorders. Whether such effects are mediated by baseline characteristics will be tested. Given suvorexant is an FDA approved treatment for insomnia, sleep will be evaluated as well in the nicotine dependent arm.

Endpoints:

In nicotine-dependent individuals, suvorexant's impact on brain function will be assessed several ways by evaluating: 1) resting function, 2) reactivity to drug cues, 3) reactivity to non-drug related cognitive tasks. Sleep and nicotine use will be measured throughout the study period. In those without nicotine-dependence, the impact of suvorexant and the interaction of acute methylphenidate and suvorexant on brain function will be assessed. This arm will provide insight into how suvorexant impacts reward/cognition as well as impacts the pharmacological influence of methylphenidate on those same measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

All Participants

* Participants will be volunteers between the ages of 18-60 at the time of enrollment in the study (both sexes). Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals.
* Participants who are able to become pregnant must have a negative pregnancy test on all study days.
* Able and willing to provide written informed consent, which includes agreement to all Lifestyle Considerations at the time of study consent.

Nicotine Dependence Arm

-Participants must be a regular smoker/vaper with a urine cotinine level corresponding to nicotine user status for the specific test being used (typically corresponding to a urine cotinine above about 200 ng/ml) and have been smoking or vaping consistently for at least the past year (excluding quit attempts).

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

All Participants

* Participants cannot meet DSM-5 criteria for lifetime and/or current psychotic disorders such as bipolar disorder, schizophrenia, schizoaffective disorder.
* Participants cannot meet DSM-5 criteria for current substance use disorders other than nicotine and marijuana and cannot meet criteria for current moderate or severe alcohol use disorder.
* Participants cannot have positive illicit drug and alcohol screen on each study visit other than for nicotine or marijuana.
* Medications with the potential to depress CNS function will be assessed by the MAI, PI, or a physician's assistant and participants excluded as necessary.
* Participants cannot have a history of major head trauma resulting in cognitive impairment, seizure, or other neurological disorders.
* Participant cannot have any history of neurological disorders, including seizures, epilepsy, or cognitive impairment which may impact MRI metrics.
* Participants cannot be pregnant or breastfeeding. Justification: The impact of suvorexant on the developing fetus and infant.
* Individuals with severe hepatic impairment will be excluded
* Participants cannot be obese as determined by a Body Mass Index (BMI) of greater than 35.
* Participants cannot be using a CYP3A inhibitor/inducer (metabolism by CYP3A is the major elimination pathway for suvorexant)
* Participants cannot have any past or present significant cardiac disorders or cerebrovascular conditions such as palpitations, tachycardia, use of the cardiac medication Digoxin, arrhythmias, acute coronary syndrome, ischemic heart disease, or uncontrolled hypertension.
* Participants cannot have narcolepsy.
* Participants cannot self-report complex sleep behaviors such as sleep driving, preparing and eating food or making phone calls.
* Participants with Major Depressive Disorder who are using medication must be stable on medication for 3 months.
* Subjects with suicidal ideation where outpatient treatment is determined unsafe.
* Subjects that cannot speak English. Justification: To include non-English speakers, we would have to translate the consent and other study documents and hire and train bilingual staff, which would require resources that we do not have and could not justify, given the small sample size for each experiment. Additionally, the data integrity of some of the cognitive tasks and standardized questionnaires used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing MRI procedures. The inability to effectively communicate MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants.
* Contraindication to MRI as determined by MRI Safety Screening form.

Nicotine Dependent Arm

* Participants cannot self-report compromised respiratory function such as severe obstructive sleep apnea or severe chronic obstructive pulmonary disease.
* Participants cannot have uncontrolled ADHD.

Control Arm

* May not have regularly used any nicotine product in the past year. Must have an expired carbon monoxide level of less than or equal to 5 ppm.
* Must not have a history of excessive substance use that may impact reward function, as evaluated by the PI, MAI, and/or designee.
* Current pharmacological treatment for opioid use disorder (i.e., use of methadone)
* May not have (or currently be treated/medicated for) any diagnoses/conditions contraindicated for use of methylphenidate.
* Participants may not have a diagnosis of ADHD (irrespective of medication use) or present with undiagnosed ADHD during screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
fMRI - cue reactivity | each scan visit
  Test whether acute and/or chronic suvorexant reduces smoking/vaping cue reactivity
cue reactivity and suvorexant effectiveness | each scan visit
  Determine whether baseline variance in cue reactivity contributes to suvorexant s effectiveness
task based fMRI | each scan visit
  Determine whether suvorexant blunts reward sensitivity
fMRI | each scan visit
  to assess not only whether there is an interaction between acute methylphenidate and suvorexant on brain function and reward/cognition, but also whether any sex differences within this interaction exist

SECONDARY OUTCOMES:
wearable watch sensor | 2 weeks of daily watch wearing
  Determine the impact of suvorexant on sleep
Resting state fMRI | each scan visit
  Determine the impact of acute and chronic suvorexant on the brain s inherent resting function

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Janes, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share data as specified in the protocol and potentially through future data transfer agreement(s). Any shared data will be stripped of identifiers prior to release for sharing. Deidentified data may be shared with properly administered databases and/or with collaborators with whom proper data sharing agreements are in place. Outside of the data sharing plan already specified in the protocol (in what would be outline in a future data sharing agreement), we have not yet finalized decisions on types of supporting information that will be shared, IPD Sharing Time Frame, IPD Sharing Access Criteria for other future data sharing agreements.